CLINICAL TRIAL: NCT03701945
Title: Pulmonary Rehabilitation Innovation and Microbiota in Exacerbations of COPD
Acronym: PRIME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Alda Sofia Pires de Dias Marques, Principal Investigator, Aveiro University
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: POCI-01-0145-FEDER-028806
Record Dates: First submitted 2018-09-25; First posted 2018-10-10 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: COPD Exacerbation; COPD
Keywords: microbiota; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: 156 patients with COPD will be followed monthly for a year and their lung microbiota and clinical data will be analysed. Community-based PR will be delivered to 56 patients. Data will be collected before, at 3 weeks, after PR and at 6 months to assess the feasibility and effects of PR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary rehabilitation (Experimental): Pulmonary rehabilitation will be provided to every patient that accepts the intervention and presents an acute exacerbation
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — Pulmonary rehabilitation will be provided to patients presenting an acute exacerbation. The intervention will be composed of exercise training, education and psychosocial support.

SUMMARY:
PRIME goal is to early detect and treat acute exacerbations of chronic obstructive pulmonary disease (AECOPD). This is important since COPD accelerates aging and represents major burden worldwide and in Portugal, mainly due to its frequent AECOPD. Pulmonary rehabilitation (PR) is an effective strategy of its management but it is scarce. When AECOPD are early detected and treated, it optimizes patients' outcomes and reduces the burden of COPD, especially if PR is used. However, up to date, there is no model to predict AECOPD for clinical practice. The lung microbiota shows promise to overcome this barrier and inform on COPD trajectory and will be investigated. In addition, despite of most AECOPD being managed in the community, PR is mainly available in hospitals and less than 1% of patients are having access. Thus, community-based PR will be implemented and a clinical decision tool developed for prioritizing who will most benefit from PR, enhancing evidence-based access to PR.

DETAILED DESCRIPTION:
PRIME aims to address these two gaps, establishing the role of microbiota and clinical data in predicting AECOPD and increasing the evidence on PR in AECOPD through the translation of PR guidelines to the community. Specifically, it aims to:

* Explore the longitudinal changes in microbiota and clinical data between stable and exacerbations periods;
* Establish the feasibility and short- and long-term effects of community-based PR for AECOPD;
* Define the characteristics of patients who most benefit from community-based PR.

  156 patients with COPD will be followed monthly for a year and their lung microbiota and clinical data will be analysed. Community-based PR will be delivered to 56 patients. Data will be collected before, at 3 weeks, after PR and at 6 months to assess the feasibility and effects of PR. A clinical decision-making tool (CDMT) to prioritise patients with AECOPD for PR will be developed.

The experienced multidisciplinary team will ensure the following novel results:

* a clinical and lung microbiota profile of patients with COPD;
* a model of AECOPD prediction;
* recommendations for community-based PR in AECOPD;
* a CDMT to prioritise patients with AECOPD for PR.

PRIME will contribute to optimise outcomes, improve AECOPD healthcare services and reduce the burden with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible if adults (≥18anos) and present a diagnose of chronic obstructive pulmonary disease (COPD).

Exclusion Criteria:

* Patients will be excluded if they had an acute cardiovascular event on the previous month or if they have a significant cardiac, immune, musculoskeletal or neurological impairment, or any other that doesn't allow them to perform tests.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in exercise tolerance | Up to 6 months
  exercise tolerance in a walking field test
Change in lung microbiota | Up to 6 months
  lung microbiota from saliva samples

SECONDARY OUTCOMES:
Change in muscle strength | Up to 6 months
  Upper and lower limb muscle strength
Change in health related Quality of life | Up to 6 months
  Measured with the St. George's Respiratory Questionnaire, that measures health related quality of life. It will be used the total score. Scores are expressed as a percentage of overall impairment where 100 represents worst possible health status and 0 indicates best possible health status.
Change in resting dyspnoea | Up to 6 months
  Resting dyspnoea measured with the modified British medical research council dyspnoea questionnaire, that ranges from 0 to 4, and is related to dyspnoea during activities of daily living. Higher scores demonstrate a higher functional impairment due to dyspnoea.
Change in self-efficacy | Up to 6 months
  self-efficacy measured with the pulmonary rehabilitation adapted index of self-efficacy tool
Change in physical activity | Up to 6 months
  Physical activity levels measured with the brief physical activity assessment tool
Change in lung function | Up to 6 months
  Lung function will be assessed through spirometry to define the airflow limitation (FEV1pp).
Change in emergency department visits | Up to 6 months
  Number of emergency visits on the previous year
Change in frequency of exacerbations | Up to 6 months
  Number of exacerbations on previous year
Change in hospitalizations | Up to 6 months
  Number of hospitalizations on previous year
Dyspnoea during exercise | Up to 6 months
  Dyspnoea experienced during exercise, monitored with the modified Borg dyspnoea scale, that ranges from 0 to 10, where 0 represents no dyspnoea and 10 the worst imaginable dyspnoea.
Fatigue during exercise | Up to 6 months
  Fatigue experienced during exercise, monitored with the modified Borg dyspnoea scale, that ranges from 0 to 10, where 0 represents no fatigue and 10 the worst fatigue the patient can imagine.

CONTACTS AND LOCATIONS:
Overall Officials: Alda Marques, PhD, Principal Investigator — School of Health Sciences, University of Aveiro
Locations (1):
- University of Aveiro, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cross AJ, Thomas D, Liang J, Abramson MJ, George J, Zairina E. Educational interventions for health professionals managing chronic obstructive pulmonary disease in primary care. Cochrane Database Syst Rev. 2022 May 6;5(5):CD012652. doi: 10.1002/14651858.CD012652.pub2. PMID 35514131